CLINICAL TRIAL: NCT02888626
Title: A Single-Center, Open-Label Pilot Study of a Novel Microlens Array Device for Skin Rejuvenation
Brief Title: Study of a Novel Microlens Array Device for Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-16-ML01
Record Dates: First submitted 2016-08-23; First posted 2016-09-05 (Estimated); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Wrinkles; Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with Microlens Array (Experimental): Treatment with Cutera Microlens Array Device used with the enlighten™ 532nm /1064nm/670nm laser
  Interventions: Device: Microlens Array

INTERVENTIONS:
Device: Microlens Array — Treatment with Cutera Microlens Array Device used with the enlighten™ 532nm /1064nm/670nm laser

SUMMARY:
A single-center prospective, open-label uncontrolled pilot study. Subjects will receive laser treatments and will be followed at 12 weeks post-final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 20 to 75 years of age (inclusive). Fitzpatrick Skin Type I - VI.
* Desires photo-rejuvenation of the skin or improvement in the appearance of acne scarring.
* Subject has visible signs of acne scarring or moderate sun-damaged and/or aging skin in the treatment area with visible areas of fine rhytides, pigmentation, erythema or telangiectasia.
* Subject must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Willing to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treatment area every day for the duration of the study, including the follow-up period.
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s), including injectable agents, for skin rejuvenation during the study and has no intention of having such procedures performed during the course of the study.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant.

Exclusion Criteria:

* Participation in a clinical trial of another drug, or device administered to the target area, within 6 months prior to enrollment or during the study.
* Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as laser or light-based procedures or surgery.
* Prior injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler within 6 months of study participation.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of retinoid, such as isotretinoin, or corticosteroid, as applicable, within 6 months of study participation.
* Topical use of retinoid, such as isotretinoin, corticosteroid or hydroquinone, as applicable, on the treatment area within 1 month of participation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — P.I.
Locations (1):
- Cutera Research Center, Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Microlens Array
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Microlens Array
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Physician's Global Assessment of Improvement
Description: Degree of improvement at 12 weeks post-final treatment as assessed by the Investigator.
  Higher scores indicate better outcomes 3= Very significant Improvement 2= Significant Improvement
  1= Moderate Improvement 0= Mild or No Improvement
Time Frame: 12 weeks post final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Microlens Array
Number analyzed (Participants) | 7
score on a scale | 2 (0.76)

ADVERSE EVENTS:
Time Frame: 12 weeks post final treatment
Arm/Group | Treatment With Microlens Array
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Microlens Array (N=7)
Erythema (Skin and subcutaneous tissue disorders) | 7
Edema (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT02888626/Prot_SAP_000.pdf